CLINICAL TRIAL: NCT00295490
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Two- Centre Study to Evaluate the Efficacy and Safety of Devil's Claw in the Treatment of Knee and Hip Osteoarthritis
Brief Title: Trial Evaluating Devil's Claw for the Treatment of Hip and Knee Osteoarthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unexpected withdrawal of funding
Sponsor: University of Southampton (Other)
Collaborators: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Principal Investigator, Dr Sarah Brien, Senior Research Fellow, University of Southampton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: devilclaw1
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: double blind randomised controlled trial; phase II; Devil's Claw; osteoarthritis of the knee; osteoarthritis of the hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Harpagophytum extract LI 174

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 240mg Devil claw (Experimental): Sub clinical dose if the 3 doses employed
  Interventions: Drug: Devil Claw
- 960mg Devil Claw (Experimental): Active dose
  Interventions: Drug: Devil Claw
- 1920 mg Devil claw (Experimental): Active dose
  Interventions: Drug: Devil Claw
- Placebo (Placebo Comparator): Comparator for all active intervention arms
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Devil Claw — Dose ranging study so will elucidate dose Frequency is four times daily
  Other Names: Harpagophytum procumbens
  Arms: 1920 mg Devil claw; 240mg Devil claw; 960mg Devil Claw
Drug: Placebo — Placebo has same dosing freq as for active intervention and for same time period
  Arms: Placebo

SUMMARY:
Osteoarthritis of both the knee and hip joints are common conditions; knee osteoarthritis affects 6% of adults over 30 years of age and osteoarthritis of the hip affects between 3% and 6% of the Caucasian population. Both forms of osteoarthritis are associated with disability. Conventional treatment (analgesics and the use non-steroidal anti-inflammatory, NSAIDS) is prophylactic, aimed at decreasing pain and improving function. However long term use of NSAIDS is associated with a high incidence of adverse events (gastrointestinal tract symptoms). A safer alternative treatment would therefore be beneficial.

Both anecdotal evidence and recent studies have implicated the potential of the herbal remedy Devil's Claw (Harpagophytum procumbens) for the treatment of painful, chronic arthritic type conditions (Ernst and Chrubasik, 2000). Devil's Claw is an extract obtained from the root of the Harpagophytum procumbens plant, a member of the sesame family found in the Kalahari region in South Africa. It has been shown that this herbal remedy has anti-inflammatory and analgesic effects (Baghdikian et al, 1997). Currently Devil's Claw is marketed for use as a supportive treatment of degenerative arthrosis, is not a Medicines Control Agency licensed product and is freely available to the general public in health food stores and pharmacies.

The objectives of this study are to assess the efficacy, optimum dosage and safety of the herbal remedy Devil's Claw (Harpagophytum) in the treatment of osteoarthritis of the knee and/or hip. The primary objective of this study is to investigate the following three principal questions:

1. To compare the efficacy of Devil's Claw with placebo in the treatment of osteoarthritis of the knee and/or hip
2. To determine the optimum dose of Devil's Claw and
3. To evaluate the safety and tolerability of three doses of Devil's Claw in the treatment of osteoarthritis of the knee/hip and to compare them to placebo There are also a number of secondary research objectives that will also be addressed (see later).

These objectives are based on the following hypotheses :

Hypotheses

* Devil's Claw has anti-inflammatory properties (as assessed by the reduction in pain, stiffness and disability aspects on the WOMAC) in chronic osteoarthritis of the knee and/or hip after 16 weeks of treatment, as compared to placebo.
* A dose response effect exists in the treatment of osteoarthritis of the knee/hip by Devil's Claw.

DETAILED DESCRIPTION:
STUDY DESIGN: Randomized, placebo-controlled, dose-ranging two-centre study PREPARATIONS FOR INVESTIGATION: Devil's Claw (Allya®)/placebo as tablets

STATISTICAL METHODS:

Analysis on an intention to treat basis.

The following tests will be performed and all statistical significance will be set at p < 0.05:

Primary efficacy analysis: The primary outcome will be the reduction in WOMAC total score from baseline to week 16. The week 16 means for the four treatment groups will be compared using an analysis of covariance taking account of baseline assessments and any demographic differences, age, gender, etc, which are found to be significant. Multiple comparison tests will be used to examine specific differences of initially specified interest, such as the two highest doses of Devil's Claw versus placebo.

Secondary Efficacy Analysis: Similar analyses of covariance will be used to examine treatment group differences at week 16 compared with baseline for WOMAC subscales (pain, stiffness and physical function), and Quality of Life assessments (SF-36). Changes in the subject's well-being and overall global assessment will be compared using appropriate non-parametric tests, e.g. Mann-Whitney test or MacNemar's test. Changes in attitudes and health beliefs to CAM will be assessed using Chi-Squared tests.

Safety Evaluation: Group differences between adverse event reporting will be assessed by descriptive methods.

NUMBER OF PATIENTS:

264 (50 patients in each group, with an expected total of 64 drop-outs) NUMBER OF SITES: 2

TIME SCHEDULE:

Study Start: April 2004 Study End: March 2007 Observation period/patient: 20 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients with either a pragmatic diagnosis of osteoarthritis of the knee, with no other known rheumatological condition and who report the following clinical features (based on the ACR classification for knee OA1):

  * knee pain on most days of the previous month
  * morning stiffness of less than 30 minutes duration
  * "stiffness" in resting the joint and and are aged over 40 years
* osteoarthritis of the hip, with no other known rheumatological condition and who report the following clinical features (based on the ACR classification for hip OA2):

  * hip pain on most days of the previous month and at least two of the following 3 features:
  * ESR < 20mm/hour
  * Radiographic femoral or acetabular osteophytes
  * Radiographic joint space narrowing (superior, axial and/or medial)
  * And are aged over 45 years of age
* The diagnosis of osteoarthritis will be confirmed by X-ray. Only patients who have grade 2 to 4 of the Kellgren and Lawrence scale will be recruited. (The Kellgren and Lawrence scale ranges from grade 0 to grade 4 where grades 0 and 1 represent doubtful osteoarthritic changes and therefore a doubtful diagnosis.)
* Patients who have been on stable medication (conventional or complementary, including nutritional medicine) for the past three months, but are still getting symptoms (incomplete responders)
* Only those patients who record baseline pain scores on the WOMAC scale of at least 20 mm on the VAS for a minimum of 6 out of 7 days monitored during the period from Clinic Visit 1 (screening) and Clinic Visit 2 (baseline)
* Ability to comply with the requirements of the study and to give informed consent
* For women of child-bearing potential: negative pregnancy test

Exclusion Criteria:

* Participation in an investigational trial within 30 days prior to enrollment
* Previous treatment with Devil' s Claw within 90 days prior to enrollment
* Patients awaiting a replacement knee or hip joint
* Patients with other conditions that cause pain
* Patients with congenital dislocation of the hip
* Patients who have had operations on their hip due to previous trauma
* Patients with severe co-morbidities - including severe cardiac or pulmonary disease and cancer
* Dementia, psychoses, or other significant impairment of mental status that would prohibit sufficient comprehension, provision of informed consent and to allow undertaking of the necessary self-care or toxicity reporting
* Patients taking corticosteroid medication
* Known allergies against any of the ingredients of the treatments
* Patients who would be unable to complete the self assessment forms, or to attend for X-ray and clinical examination
* Patients with other known rheumatic disease such as rheumatoid arthritis
* Patients with the diagnosis gout
* Patients who report a red or hot swollen joint (which is unlikely to be due to OA), and would require further rheumatological assessment
* Patients with conditions known to be contraindicated to the study medication i.e. patients with gastric or duodenal ulcers; gallstones; patients taking drugs for arrhythmias; patients with heart failure
* Patients who are pregnant, trying to become pregnant or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-12; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Lewith, MA MD FRCP, Principal Investigator — University of Southampton; Sarah Brien, Bsc Msc PhD, Principal Investigator — University of Southampton
Locations (1):
- Wellcome Trust Clinical Research Facility, Southampton General Hospital, Southampton, Hants, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited during 2004 to 2007 Recruitment location: From GP clinics and from adverts in the media
Pre-assignment Details: Patients attended screening clinic to confirm diagnosis of osteoarthritis of the knee (grade 2-4) by clinical examination and X ray and ensure other entry criteria met i.e.baseline pain (at least 20mm on 100mm scale over 6 of 7 days between screening and baseline)and exclude any other condition causing knee pain.
Groups:
- 240mg Devil Claw: Total daily dose was 240mg/day taken orally; this dose is suboptimal. Patients allocated to this treatment arm receiving eight tablets split into two doses to take daily for 16 weeks. of these eight tablets, 7 were placebo medication and one was active Devil Claw (the active tablet contained 240mg Devil Claw).
- 960mg/d Devil Claw: total daily dose was 960mg/day taken orally. Patients allocated to this treatment arm receiving eight tablets split into two doses to take daily for 16 weeks. of these eight tablets, 4 were placebo medication and four were active Devil Claw, with each active tablet containing 240mg Devil Claw .
- 1,920mg/d Devil Claw: total daily dose was 1920mg/day of Devil claw taken orally. Patients allocated to this treatment arm receiving eight tablets split into two doses to take daily for 16 weeks. All eight tablets contained active Devil Claw; each active tablet containing 240mg Devil Claw .
- Placebo: total daily dose was 0mg/day of Devil Claw. Patients allocated to this treatment arm receiving eight tablets split into two doses to take daily for 16 weeks. of these eight tablets, all were placebo medication. tablets were taken orally.
Period: Overall Study
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Started | 15 | 19 | 16 | 17
Completed | 14 | 15 | 12 | 12
Not Completed | 1 | 4 | 4 | 5
Not completed — Protocol Violation | 0 | 0 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo | Total
Number analyzed (Participants) | 15 | 19 | 16 | 17 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 13 | 11 | 9 | 39
  >=65 years | 9 | 6 | 5 | 8 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (11.9) | 59.6 (6.9) | 59.8 (8.4) | 63.2 (8.6) | 61.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 8 | 9 | 32
  Male | 10 | 9 | 8 | 8 | 35
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 19 | 16 | 17 | 67

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and Mc Master University OA Index (WOMAC)
Description: WOMAC is a disease specific outcome measure for osteoarthritis. It has three subscales assessing pain (5 questions), stiffness (2 questions) and function (15 questions). together the subscales give an overall total score ranging from 0 (worst) to 100 (best; an increase in total score indicates an improvement in health. THe outcome was measured at baseline, week 8 and week 16. In this study the primary outcome was the reduction in WOMAC total score from baseline to the end of treatment at week 16.
Time Frame: Baseline, week 8 and week 16
Population: Zero participants were analysed as the study was terminated prematurely.
Measure: Mean (Standard Deviation); unit: Unit on 100mm scale
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Pain Subscale on Western Ontario and Mc Master University OA Index
Description: Subscale assessed by 100mm VAS based on five questions addressing pain in osteoarthritis using the terminators no pain (0mm) to extreme pain (100mm). a higher score therefore indicates more severe pain. This outcome was recorded at baseline, week 8 and week 16 (end of treatment). The outcome for this study was reported as the change in WOMAC pain score from baseline to end of treatment at week 16.
Time Frame: Baseline, week 8 and week 16
Population: Zero participants were analysed as the study was terminated prematurely.
Measure: Mean (95% Confidence Interval); unit: Unit on 100mm VAS scale
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Disability Subscale on The Western Ontario and Mc Master University OA Index
Description: Subscale assessed by 100mm VAS based on twelve questions addressing disability in osteoarthritis with a higher score indicating worse symptoms. The VAS used terminators of no disability (0mm) to extreme disability (100mm). The measure was recorded at baseline, week 8 and week 16. We reported the outcome as the change from baseline to end of treatment at week 16.
Time Frame: baseline, 8 and 16 weeks
Population: Zero participants were analysed as the study was terminated prematurely
Measure: Mean (95% Confidence Interval); unit: unit on 100mm VAS scale
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Stiffness Subscale on the The Western Ontario and Mc Master University OA Index
Description: Subscale assessed by 100mm VAS based on two questions addressing stiffness in osteoarthritis;a higher score indicating worse symptoms. The VAS used terminators of no stiffness (0mm) to extreme stiffness (100mm). The measure was recorded at baseline, week 8 and week 16. We reported the outcome as the change from baseline to end of treatment at week 16.
Time Frame: Baseline, week 8 and week 16
Population: Zero participants were analysed as the study was terminated prematurely.
Measure: Mean (95% Confidence Interval); unit: Unit on 100mm VAS scale
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Short Form-36 (SF-36)
Description: Quality of Life assessment containing 8 scales clustered into 2 summary scales: physical health and mental health. Each question is scored out from 0 (indicating worst health) to 100 (indicating best health). Mean scores for the 8 scales (total scores/no questions completed) are calculated to give a total score for each of the two summary scales between 0 (worst health) and 100 (best health). SF36 was recorded at baseline, week 8 and at the end of treatment at week 16. we reported the change from baseline to end of treatment as the outcome.
Time Frame: Baseline, week 8 and week 16
Population: Zero participants were analysed as the study was terminated prematurely.
Measure: Mean (95% Confidence Interval); unit: Unit of scale
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Patient Global Assessment
Description: To assess changes in the subject's well-being based on 7 point likert scale ranging from very poor (0 point) to very good (7 point). Outcome was recorded at baseline, week 8 and end of treatment at week 16. We reported outcome as the change in patient global assessment from baseline to end of treatment at week 16.
Time Frame: Baseline, week 8 and week 16
Population: Zero participants were analysed as the study was terminated prematurely
Measure: Mean (95% Confidence Interval); unit: Unit on scale (Likert from very poor to
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Complementary and Alternative Medicine Beliefs Inventory
Description: Questionnaire to assess changes in attitudes and health beliefs to CAM.the questionnaire as 17 questions, each scored on a 7 point likert scale from strongly disagree to strongly agree; a higher score indicates stronger belief in the measure. Minimum score 17, maximum score 119
Time Frame: four monthly
Population: Zero participants were analysed as the study was terminated prematurely
Measure: Mean (95% Confidence Interval); unit: unit on scale
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Adverse Event Reporting
Description: To identify Group differences between the number of adverse event recorded by patient for both serious and non serious adverse events, as well as events considered being attributable to the study medication.
Time Frame: Baseline and weeks 2,4,6,8,12 and 16
Population: Zero participants were analysed as the study was terminated prematurely
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Twenty week period
Arm/Group | 240mg Devil Claw | 960mg/d Devil Claw | 1,920mg/d Devil Claw | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/19 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 15/15 | 18/19 | 15/16 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240mg Devil Claw (N=15) | 960mg/d Devil Claw (N=19) | 1,920mg/d Devil Claw (N=16) | Placebo (N=17)
Transient blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 240mg Devil Claw (N=15) | 960mg/d Devil Claw (N=19) | 1,920mg/d Devil Claw (N=16) | Placebo (N=17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 11 (11) | 9 (9) | 11 (11)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 2 (2) | 2 (2)
Headache (General disorders) | 5 (5) | 5 (5) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes